CLINICAL TRIAL: NCT06433466
Title: The Impact of Instagram and TikTok Influencer Marketing on Perceptions of E-cigarettes in Young Adults: a Survey-based Experiment
Brief Title: Influencer Marketing: a Survey-based Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jennifer Unger, Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: unidentified
Record Dates: First submitted 2024-05-14; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videos featuring influencers promoting e-cigarettes alongside healthy lifestyle activities (Experimental): Young adults were randomly shown 10 videos, featuring influencers promoting e-cigarettes alongside healthy lifestyle activities (experimental group).
  Interventions: Other: Videos featuring influencers promoting e-cigarettes alongside healthy lifestyle activities
- Videos featuring influencers showing healthy lifestyle activities (Active Comparator): Young adults were randomly shown 10 videos, featuring influencers promoting healthy lifestyle activity alone (control).
  Interventions: Other: Videos featuring influencers promoting e-cigarettes alongside healthy lifestyle activities

INTERVENTIONS:
Other: Videos featuring influencers promoting e-cigarettes alongside healthy lifestyle activities — Young adults were randomly shown 10 videos, featuring influencers promoting e-cigarettes alongside healthy lifestyle activities (experimental group), or a healthy lifestyle activity alone (control).

SUMMARY:
Young adults (N = 1,500) will participate in the online survey-based experiment. They will be randomly shown 10 videos, featuring influencers promoting e-cigarettes alongside healthy lifestyle activities (experimental group), or a healthy lifestyle activity alone (control). After watching each video, participants will rate perceptions of influencer credibility (i.e., honesty, trustworthiness, knowledge, attractiveness, intelligence, and popularity) on the scale of 0 (e.g., dishonest) to 100 (honest).

Among all participants, harm perceptions of e-cigarettes will be assessed. Susceptibility to use e-cigarettes will be assessed among never users. These outcomes will then be compared among participants who perceived influencers as credible and those who perceived influencers as non-credible.

DETAILED DESCRIPTION:
Young adults (18-24 years of age) living in California were recruited by YouGov marketing research panel to participate in a survey on tobacco-related attitudes and behaviors. YouGov, a research panel agency, has been used in prior research to survey young adults about their tobacco-related attitudes and behaviors. Respondents (N=1,500) were matched to a sampling frame based on gender, age, race, and education. The sampling frame was a politically representative modeled frame of United States (U.S.) adults based on the American Community Survey. The matched cases were weighted to the sampling frame using a propensity score matching procedure. Participants were provided with a survey URL link. After completing informed consent, participants completed the survey online. The study was approved by the University of Southern California Institutional Review Board (UP-21-00135). Respondents were randomly assigned to watch 10 10-second long TikTok videos in either experimental (influencers promoting e-cigarettes alongside healthy lifestyle activities ) or control group (influencers showing healthy lifestyle activity alone).

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years of age,
* English fluency,
* Current California resident.

The survey was sampled to be representative by age group (18 to 24) and gender, and was weighted to be representative by age, gender, race, and educational attainment using propensity score weighting.

Exclusion Criteria:

Not meeting these criteria:

* 18-24 years of age,
* English fluency,
* Current California resident.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1500 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
harm perceptions of e-cigarettes | one-time assessment after the experimental exposure (immediately post-treatment)
  Responses to the question, "Do you think vaping e-cigarettes is harmful to your health?" were measured on a Likert scale, ranging from "definitely yes" (1), "probably yes" (2), to "probably not (3)," "definitely not (4)." The measure represents one validated item from the Population Assessment of Tobacco and Health (PATH).
Susceptibility to use e-cigarettes | one-time assessment after the experimental exposure (immediately post-treatment)
  Susceptibility to use e-cigarettes was measured (among never-users of e-cigarettes), using the validated three-item scale adapted from PATH, and combined into one variable (α=0.93). Consistent with prior research, the measure was dichotomized with responses "definitely not" to all items being coded as "not susceptible" and responses "probably not," "probably yes", or "definitely yes" being coded as "susceptible."
Perceptions of influencer credibility | assessed 10 times after each video (during treatment, immediately after each video)
  Perceptions of influencer credibility (i.e., honesty, trustworthiness, knowledge, intelligence, attractiveness, and popularity) were assessed using a 0 (e.g., dishonest) -100 (e.g., honest) scale that has been validated in prior research.

CONTACTS AND LOCATIONS:
Locations (1):
- YouGov, online, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vassey J, Vogel EA, Unger JB, Cho J, Bae D, Donaldson SI, Allem JP. Impact of Instagram and TikTok influencer marketing on perceptions of e-cigarettes and perceptions of influencers in young adults: a randomised survey-based experiment. Tob Control. 2025 Feb 13:tc-2024-059021. doi: 10.1136/tc-2024-059021. Online ahead of print. PMID 39947698